CLINICAL TRIAL: NCT07131748
Title: Effect of Heated Water-Based Versus Land-Based Exercise Training on Hemodynamic Variables, Functional Capacity and Quality of Life in Older
Brief Title: Effect of Heated Water-Based Versus Land-Based Exercise Training on Hemodynamic Variables, Functional Capacity and Quality of Life in Older Hypertensive
Acronym: HExOLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Emmanuel Gomes Ciolac, Associate Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017/25648-4
Record Dates: First submitted 2019-10-24; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Aging; Exercise
Keywords: Aging; Exercise; Pathophysiology; Hypertension; Elderly; Hemodynamic Response
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Intervention Model Description: HAS HEX vs HAS LEX HAS HEX vs HAS CON HAS LEX vs HAS CON
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HAS HEX vs HAS LEX (Experimental)
  Interventions: Other: Physical Exercise Session in heated Swimming Pool - HEx; Other: Physical Exercise Session in Land- LEx
- HAS HEX vs HAS CON (Experimental)
  Interventions: Other: Physical Exercise Session in heated Swimming Pool - HEx; Other: Control Session Without Exercise- CON
- HAS LEX vs HAS CON (Experimental)
  Interventions: Other: Physical Exercise Session in heated Swimming Pool - HEx; Other: Control Session Without Exercise- CON

INTERVENTIONS:
Other: Physical Exercise Session in heated Swimming Pool - HEx — Warm Up - 5 minutes of stretching and heating of the joints and muscle groups to be worked; Aerobic exercise - 30 minutes of aerobic exercise (following the same control parameter of the experimental session); Resistance exercises - 20 minutes of resisted exercises, which will be divided into 6 exercises with 2 sets of 10 to 15 repetitions (following the same control parameter of the experimental session); Calm back - 5 minutes of stretching.
Other: Physical Exercise Session in Land- LEx — Warm up - 5 minutes of stretching and heating of the joints and muscle groups to be worked; Aerobic exercise - 30 minutes of aerobic exercise performed on treadmill and / or exercise bike (following the same control parameter of the experimental session); Endurance Exercises - 20 minutes of exercises resisted, also divided into 6 exercises with 2 sets of 10 to 15 repetitions. The large muscle groups of the upper limbs, lower limbs and trunk will be exercised in fitness machine and with free weights (following the same control parameter of the experimental session); Calm back - 5 minutes of stretching.
  Arms: HAS HEX vs HAS LEX
Other: Control Session Without Exercise- CON — Guidance to maintain the usual level of physical activity and not to enter physical exercise programs during the 12 weeks of follow-up.
  Arms: HAS HEX vs HAS CON; HAS LEX vs HAS CON

SUMMARY:
BACKGROUND: Physical exercise promotion is one of the main global goals of innumerous health and medical societies for preventing and managing noncommunicable chronic diseases (NCDs), being one of the main therapeutic for the patient with hypertension. Exercise in heated swimming pool has emerged as a potential alternative to physical exercise on the ground for the reduction of blood pressure (BP) of hypertensive patients, however, its effects on BP, as well as hemodynamic, metabolic, inflammatory and functional variables of older individuals with hypertension have not been investigated.

PURPOSE: To evaluate the effects of heated water-based exercise (HEx) versus land-based exercise (LEx) on BP, arterial stiffness, endothelial function, metabolic, inflammatory and functional variables of older individuals with hypertension.

METHODS: 60 older individuals (male and female) with hypertension (age > 60 years) will be randomized in 2:2:1 ratio to HEx, LEx or control (CON) intervention. The feasibility and physiological adaptations (physical capacity, musculoskeletal and cardiovascular responses to stress, biological and biochemical markers associated with the pathophysiology of the disease and vascular adaptations) will be assessed before, after 12 weeks and after 24 weeks of follow-up. HEx and LEx training programs will be performed three times per week and will be performed for the firs 12 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

- For the study population, the following will not be included in the study:

* Smokers (avoiding acute effects of smoking on physiological measures);
* Individuals with decompensated cardiovascular disease, thyroid dysfunction and / or inflammatory diseases;
* Unable individuals to perform an exercise program or ergospirometric test due to physical or mental incapacity;
* Individuals with hemodynamic and / or electrocardiographic changes during the ergospirometric test.
* Only individuals older than 60 years, with a diagnosis of SAH for more than 6 months (stage 1 or 2), using antihypertensive medication (office BP less than 140/90 mmHg) and without medication change for at least 2 months.

Exclusion Criteria:

* For the study population, individuals who have less than 60% adherence to scheduled physical exercise sessions will be excluded during the study.
* Individuals who change or discontinue their clinical and / or pharmacological treatment (with or without a prescription).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure change | baseline, 3 month and 6 month
  24-hour systolic and diastolic ambulatory blood pressure change from baseline

SECONDARY OUTCOMES:
Arterial stiffness | baseline, 3 month and 6 month
  Carotid-femoral pulse wave velocity change from baseline
Brachial artery flow-mediated dilation (FMD) | baseline, 3 month and 6 month
  Change from baseline in brachial artery flow-mediated dilation (FMD) (%), calculated as: (peak diameter - baseline diameter) / baseline diameter × 100, measured via ultrasound (SonoSite M-Turbo™) after 5-minute artery occlusion.
Maximal oxygen consumption | baseline, 3 month and 6 month
  Change from baseline of maximal oxygen consumption during a progressive cardiopulmonary exercise testing
First ventilatory threshold (anaerobic threshold) | baseline, 3 month and 6 month
  Change from baseline in the first ventilatory threshold (anaerobic threshold) will be measured by the V-slope method during a progressive cardiopulmonary exercise testing.
Change from baseline in the second ventilatory threshold (respiratory compensation point) | baseline, 3 month and 6 month
  Change from baseline in the second ventilatory threshold (respiratory compensation point) will be determined determined as the point at which a rapid rise in ventilation/carbon dioxide output, and a fall in partial pressure of carbon dioxide output during a progressive cardiopulmonary exercise testing.
Exercise tolerance | baseline, 3 month and 6 month
  Change from baseline of exercie duration (minutes) during a progressive cardiopulmonary exercise testing
Handgrip strength | baseline, 3 month and 6 month
  Change from baseline of maximum isometric strength measured during handgrip strength testing (dynamometry)
Flexibility | baseline, 3 month and 6 month
  Change from baseline of the seat-and-reach test performance
Lower-limb strength | baseline, 3 month and 6 month
  Change from baseline of the five time sit-to stand performance
Agility and balance | baseline, 3 month and 6 month
  Change from baseline of the timed-up and go test performance
Endurance performance | baseline, 3 month and 6 month
  Six-minute walking test performance change from baseline

OTHER OUTCOMES:
Interleukin 6 | baseline, 3 month and 6 month
  Change from baseline of plasma levels of Interleukin 6
C-reactive protein | baseline, 3 month and 6 month
  Change from baseline of plasma levels of C-reactive

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Estadual Paulista Julio de Mesquita Filho, Bauru, São Paulo, Brazil